CLINICAL TRIAL: NCT02536417
Title: Efficacy of Melatonin in Decreasing the Incidence of Delirium in End of Life Patients: A Randomized Double-blinded Placebo Controlled Pilot Study
Brief Title: Efficacy of Melatonin in Decreasing the Incidence of Delirium in End of Life Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fraser Health (Other)
Responsible Party: Principal Investigator, David Ng, Clinical Pharmacy Specialist, Fraser Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FHREB 2015-048
Record Dates: First submitted 2015-08-10; First posted 2015-08-31 (Estimated); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Delirium
Keywords: Melatonin; Delirium prevention; End-of-life
MeSH Terms: conditions — Delirium; Death | interventions — Melatonin; Sugars; Lactose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Treatment arm: melatonin (Active Comparator): melatonin 0.5 mg as treatment, to be given daily at bedtime
  Interventions: Drug: Melatonin
- Placebo arm (Placebo Comparator): Sugar pill identical in appearance to the melatonin 0.5 mg tablets used in treatment arm
  Interventions: Drug: Sugar pill

INTERVENTIONS:
Drug: Melatonin — To determine the effectiveness of melatonin in preventing the development of delirium compared with placebo
  Other Names: Melatonin Brand: General Nutrition Center
  Arms: Treatment arm: melatonin
Drug: Sugar pill — To determine if placebo effect plays a part in preventing the development of delirium
  Other Names: Lactose pill
  Arms: Placebo arm

SUMMARY:
The purpose of this study is to determine if melatonin administration to end-of-life patients is effective in preventing the development of delirium compared with those who do not receive this treatment. Delirium is a difficult to control symptom commonly seen in patients at the end-of-life. A person who is delirious is unable to think clearly and cannot make sense of what is going on around him/her.

DETAILED DESCRIPTION:
All patients over the age of 19 admitted to the tertiary palliative care unit and hospice residence who could meet the study requirements will be asked within 48 hours of admission for their interest in participating in the study. All those who interested in taking part will be referred to a research nurse for initial assessment for eligibility. For eligible patients who have consented to participate in the study, a research nurse who is not directly involved in the patient's care will approach the patient. A detailed subject information containing pertinent information on the study will be provided and ample time (up to 24 hours) will be given for consideration. The research nurse will explain the consent form to the patient and obtain consent signature if he/she agrees to participate. Once formal consent obtained, the eligible patient will be enrolled in the study.

Patients will be assigned randomly to one of the two arms of the study and receive nightly doses of melatonin 0.5 mg or placebo. Patients will be monitored for 14 days or until the development of delirium or the occurrence of death.

Patients will be assessed twice a day for delirium, around the end of each nursing shift, i.e. every 12 hours (at 0330 & 1530h) for fourteen consecutive days or until the development of delirium. The diagnostic tool used to detect delirium is the Confusion Assessment Method (CAM).

The primary outcome measure is incidence of delirium, defined according to the Confusion Assessment Method (CAM).

Data on harm will be collected. For example, adverse effects from melatonin such as excessive daytime drowsiness, headaches, nausea , transient depression have been reported in the medical literature. Patients will also be monitored closely for the development any of these adverse effects during the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the test site
* Adult patients over 19 years of age
* Patients who can provide informed consent
* Patients who are able to tolerate oral medications

Exclusion Criteria:

* Patients with existing delirium or dementia on admission
* Patients with poor clinical performance
* Patients taking melatonin prior to admission
* Patients taking medications that interact with melatonin
* Patients who are unable to provide informed consent
* Patients who are enrolled in any other research study involving drugs/devices

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-06-29 (Actual); Primary Completion 2020-09 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Development of delirium, as determined by the Confusion Assessment Method (CAM) criteria | 1 month
  The CAM diagnostic scale is a diagnostic instrument for identification of delirium for use in alert, non-intubated patients . It is a widely accepted and reliable tool for the detection of delirium in multiple clinical and research settings. The CAM method detects delirium using four key delirium criteria: (a) acute mental status change, (b) inattention, (c) disorganized thinking, and (d) altered level of consciousness. Delirium is diagnosed when criteria (a) and (b) plus either (c) or (d) are present.

CONTACTS AND LOCATIONS:
Overall Officials: David D Ng, PharmD, Principal Investigator — Fraser Health
Locations (1):
- Surrey Memorial Hospital, Surrey, British Columbia, Canada